CLINICAL TRIAL: NCT05128305
Title: Shandong Provincial Integrated Traditional Chinese and Clinical Medicine(Chronic Hepatitis B and Its Complication) Prevention and Treatment Project
Brief Title: Integrated Traditional Chinese and Clinical Medicine for Chronic Hepatitis B and Its Complication
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Lili Cao, Professor, Qianfoshan Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-2020-1230
Record Dates: First submitted 2021-10-10; First posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Hepatic Encephalopathy; Cirrhosis, Liver; Portosystemic Shunt
MeSH Terms: conditions — Hepatic Encephalopathy; Liver Cirrhosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group 1 (Experimental): traditional chinese medicine 1 and traditional chinese medicine 2 simulant
  Interventions: Drug: traditional Chinese medicine1 and traditional Chinese medicine 2
- group 2 (Experimental): traditional chinese medicine 1 simulant and traditional chinese medicine 2
  Interventions: Drug: traditional Chinese medicine1 and traditional Chinese medicine 2
- group 3 (Experimental): traditional chinese medicine 1 and traditional chinese medicine 2
  Interventions: Drug: traditional Chinese medicine1 and traditional Chinese medicine 2
- group 4 (Placebo Comparator): traditional chinese medicine 1 simulant and traditional chinese medicine 2 simulant
  Interventions: Drug: traditional Chinese medicine1 and traditional Chinese medicine 2

INTERVENTIONS:
Drug: traditional Chinese medicine1 and traditional Chinese medicine 2 — We use two traditional Chinese medicine prescriptions to intervene in patients after TIPS
  Other Names: traditional Chinese medicine1 simulant and traditional Chinese medicine 2 simulant

SUMMARY:
Hepatic encephalopathy is the most common complication after TIPS, and hepatic encephalopathy occurs in almost all portosystemic shunts. For patients with severe upper gastrointestinal bleeding or refractory ascites in the decompensated chronic hepatitis B, transjugular intrahepatic portosystemic shunt (TIPS) is a very effective treatment. However, due to the severe complications such as hepatic encephalopathy after TIPS, the clinical application of TIPS is limited. Literature studies have shown that the incidence of encephalopathy after TIPS is about 35%. TIPS reduces the portal vena blood flow into the liver by establishing a new channel. But at the same time, the toxic substances from the gastrointestinal tract and other organs do not enter the liver to detoxify, and are more likely to enter the brain, leading to hepatic encephalopathy.

Moreover, studies have found that the liver and the intestine originate from the same germ layer and are closely related to each other in anatomy and function. There are a large number of microorganisms living in the intestinal tract. Normally, the intestinal tract, as the first defense of the human body, can effectively prevent bacteria and their products from entering the bloodstream. In cirrhosis and portal hypertension, blood return disorder causes intestinal damage. A series of microbes and product endotoxins such as gram-negative bacteria will enter the blood through the injury, and the toxins in the peripheral blood will enter the brain and cause hepatic encephalopathy happened.

The research team's early treatment plan with integrated traditional Chinese and Western medicine proved that it greatly reduced the incidence of hepatic encephalopathy after TIPS. And improve the clinical symptoms and signs of patients with liver cirrhosis, and improve the quality of life and survival of patients.

ELIGIBILITY:
Inclusion Criteria:

* TIPS treatment criteria in line with the 2017 edition of the "Expert Consensus on Transjugular Intrahepatic Portosystemic Shunt" were selected to include patients with hepatitis B cirrhosis and Child-pugh grade A and B after TIPS surgery.
* Patients with liver cirrhosis, portal hypertension, bleeding from esophagus and gastric varices; refractory pleural and ascites due to liver cirrhosis; incomplete portal vein/localized thrombosis in liver cirrhosis or primary and secondary prevention of cirrhosis, portal hypertension, esophagus and gastric varices bleeding.

Exclusion Criteria:

* Severe blood coagulation disorder (PTA≤20%) or platelets lower than 30×109/L;
* Child-pugh classification of liver function C;
* Those with respiratory and circulatory dysfunction;
* Those whose systemic or focal infections have not been effectively controlled;
* Patients with moderate to severe malnutrition;
* Extensive primary or metastatic liver malignant tumors;
* Those who are highly allergic to the products and drugs used in the treatment process.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of hepatic encephalopathy | 12 weeks of treatment
  The incidence of hepatic encephalopathy after 12 weeks of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- he First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital, Jinan, Shandong, China